CLINICAL TRIAL: NCT03466216
Title: A Phase 1, Non-Randomized, Open-Label, Dose Escalation, Single-Center Study to Determine the Safety, Bio-distribution, and Preliminary Effectiveness of AlphaMedix™ in Adult Subjects With SSRT(+) NETs.
Brief Title: Phase 1 Study of AlphaMedix™ in Adult Subjects With SSTR (+) NET
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated for non-safety reasons.
Sponsor: Orano Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALPHAMEDIX01
Record Dates: First submitted 2018-01-11; First posted 2018-03-15 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Neuroendocrine Tumor
Keywords: somatostatin receptor
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AlphaMedix (Experimental): There is only a single treatment arm.
  Interventions: Drug: AlphaMedix

INTERVENTIONS:
Drug: AlphaMedix — There is only a single treatment intervention.
  Other Names: Pb212-octreotide analog

SUMMARY:
AlphaMedix™ (²¹²Pb-DOTAMTATE) is a radiotherapeutic drug indicated in subjects with unresectable, metastatic somatostatin receptor (SSTR) positive neuroendocrine tumors (NETs). Because 212Pb is an in vivo generator of alpha particles, it is particularly suitable for SSTR therapy applications.

This drug addresses an unmet need in the field of peptide receptor radionuclide therapy (PRRT) for NETs. Substitution of an alpha emitter (²¹²Pb) for the beta emitters currently being used (i.e., 177Lu or 90Y) will provide significantly higher Linear Energy Transfer (LET) and a shorter path length. Higher LET particles should cause more tumor cell death. Shorter path length should result in less collateral damage of the normal tissue and therefore less side effects for subjects receiving the drug.

DETAILED DESCRIPTION:
This dose escalation study will include a maximum of 50 subjects with histologically confirmed NET, a positive somatostatin analogue scan, and no prior history of PRRT therapy.

The study will begin with a single ascending dose (SAD) of AlphaMedix™ administered by IV. Subsequent cohorts will receive an incremental 30% increase that will continue until tumor response or DLT. Once tumor response is observed, the study will convert to a Multiple Ascending Dose (MAD) regimen. The MAD treatment regimen will start with the previous safe cohort's dose and will consist of 3 IV administrations of AlphaMedix™ at 8-week intervals. Subsequent cohorts will receive an incremental 30% increase that will continue until tumor response or DLT.

The primary objective is to assess the safety and dose limiting toxicity (DLT) using ascending doses of AlphaMedix™. The secondary objectives are to determine the pharmacokinetic properties and preliminary effectiveness of AlphaMedix™.

ELIGIBILITY:
Inclusion Criteria:

* ECOG status 0-2.
* Life expectancy of at least 12 weeks.
* Histologically confirmed diagnosis of SSTR (+) NET, unresectable or metastatic.
* Measurable disease per RECIST 1.1 on CT/MRI scans, defined as at least 1 lesion with ≥ 1 cm in longest diameter (LD) (lymph nodes along short axis).
* Appropriate diagnostic imaging studies, at the discretion of the PI including but not limited to CT, MRI, 18F-FDG PET/CT, NAF PET/CT bone scan, ultrasound, etc. of the tumor region or suspected area within the 4 weeks of dosing day.
* SSTR(+) disease, as evidenced by available FDA approved SSTR imaging (SRI) within 4 weeks prior to the first cycle.
* All FDA-approved therapies for which the subject is eligible have been exhausted.
* Recent blood test results (within 2 weeks pre-dose) as follows: Sufficient bone marrow capacity as defined by white blood cell (WBC) ≥2,500/µl and WBC ≥2,000/µl for subsequent cycles; platelets ≥ 100,000/µl for the first treatment and ≥75,000 for the subsequent therapies, hemoglobin (HgB) ≥8.9 g/dl for the first treatment and 8.0 g/dl for the subsequent therapies, ANC ≥1,500/µl for the first treatment and ≥1,000/µl; for the subsequent therapies; ALT, AST values ≤3 times upper limit of normal (ULN); Bilirubin: ≤3 times ULN; Serum creatinine ≤150 µmol/liter or 1.7 mg/dl; Negative pregnancy test in women capable of child-bearing within 48 hours of administration; Serum albumin > 3.0 g/L (<3.0 g/L may be acceptable at the discretion of PI, if PT, PTT, and INR are within normal range)

Exclusion Criteria:

* Prior whole-body radiotherapy and PRRT using 177Lu/90Y/111In- DOTATATE/DOTATOC or TAT
* Known hypersensitivity to 68Gallium, Octreotate, or any of the excipients of 68Ga-DOTATATE, AA infusion or AlphaMedix™.
* Therapeutic use of any somatostatin analogue, including Sandostatin® LAR (within 28 days) and Sandostatin® (within 1 day) prior to administration of investigational drug.
* Subjects with unusual hematological parameters, including an increased mean corpuscular volume (MCV) (>100,000), and especially in those who had previous chemotherapy, the advice of a hematologist should be sought for adequate further work-up to rule out myelodysplastic syndrome (MDS).
* Any subject who is taking concomitant medications that decrease renal function (such as aminoglycoside antibiotics).
* Female subjects who are pregnant, lactating or women of childbearing potential not willing to practice effective contraceptive techniques during the study period and for 8 weeks post-injection or male subjects who have female partners of childbearing potential not willing to practice abstinence or effective contraception, during the study period and for 8 weeks post-injection.
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Indication for surgical lesion removal with curative potential
* Known brain metastases; unless these metastases have been treated and stabilized 6 months prior to enrollment
* Completion of: (1) cytotoxic chemotherapy for less than 6 weeks; (2) a biological agent for less than 5 half-lives; and (3) radiation therapy for less than 6 weeks prior to study enrolment,
* Uncontrolled congestive heart failure; subjects suspected of having this condition need to show ejection fraction of >55% as determined by multigated acquisition (MUGA) scan.
* Carcinoid heart disease: Prior history of torsade de pointe, or congenital long QT syndrome; Conditions with screening ECG repolarization difficult to interpret, or showing significant abnormalities. This includes, but is not limited to: high degree AV block, pacemaker, atrial fibrillation or flutter; QTcF interval > 480 msec on screening ECG; Significant hypokalemia at screening (Potassium <3.5 mMol/L); Significant hypomagnesemia at screening (Mg++ <0.7 mMol/L)
* GFR < 35 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
To determine dose-limiting toxicity (DLT) | 8 weeks post-injection
  DLT is defined as non-hematological toxicity - all Grade 4 and Grade 3 (except alk. phos.) that is not responsive to NMT 72 hours of supportive care - and all hematological toxicity that does not recover to NMT than Grade 2 within 8 wks of dose administration.
Incidence of treatment-emergent AEs and SAEs as assessed by CTCAE v. 4 | 32 months after enrollment
  AEs will be recorded both spontaneously by the patient during the treatment period and at all safety follow ups (2 wks, 4 wks, 6 wks, 8 wks post each injection and 3 mo, 6 mo, 10 mo, 12 mo, 15 mo, 18 mo, 21 mo, and 24 mo post last injection)

SECONDARY OUTCOMES:
Partial or complete response assessed by modified RECIST v1.1 | 32 months after enrollment
  CT/MRI or 18FDG-PET/CT (for patients who are FDG-avid at baseline) will be used to measure tumor size
To determine effective blood clearance and cumulative blood activity of 212-Pb | 24 hours post-injection
  Blood will be taken at Time 0, 1 hr, 4 hr and 24 hr post-injection and measured for activity in an auto gamma counter
To determine the rate and extent of 212-Pb elimination in urine | 24 hours post-injection
  Bladder will be emptied just prior to injection and qualitative urine collections will be done 0-1 hr, 1-4 hr and 4-24 hr post-injection and measured for activity in an auto gamma counter

CONTACTS AND LOCATIONS:
Locations (1):
- Excel Diagnostics and Nuclear Oncology Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided